CLINICAL TRIAL: NCT02563847
Title: Effect of Amino Acids and Sugar Alcohols on Gastric Emptying and Release of Satiation Peptides in Normal Weight and Obese Subjects
Brief Title: Effect of Amino Acids and Sugar Alcohols on Gastric Emptying and Release of Satiation Peptides in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: EKBB 2014/072
Record Dates: First submitted 2015-05-26; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Endocrine System Diseases
MeSH Terms: conditions — Endocrine System Diseases | interventions — Tryptophan; Leucine; Xylitol; Erythritol; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- 0.52 g L-Tryptophan (Active Comparator): 0.52 g L-Tryptophan in 300 mL tap water (plus 50 mg 13C-sodium acetate) given via nasogastric tube
  Interventions: Dietary Supplement: 0.52 g L-Tryptophan; Other: 50 mg 13C-sodium acetate
- 1.56 g L-Tryptophan (Active Comparator): 1.56 g L-Tryptophan in 300 mL tap water (plus 50 mg 13C-sodium acetate) given via nasogastric tube
  Interventions: Dietary Supplement: 1.56 g L-Tryptophan; Other: 50 mg 13C-sodium acetate
- 1.56 g L-Leucine (Active Comparator): 1.56 g L-Leucine in 300 mL tap water (plus 50 mg 13C-sodium acetate) given via nasogastric tube
  Interventions: Dietary Supplement: 1.56 g L-Leucine; Other: 50 mg 13C-sodium acetate
- 50 g Xylitol (Active Comparator): 50 g Xylitol in 300 mL tap water (plus 50 mg 13C-sodium acetate) given via nasogastric tube
  Interventions: Dietary Supplement: 50 g Xylitol; Other: 50 mg 13C-sodium acetate
- 75 g Erythritol (Active Comparator): 75 g Erythritol in 300 mL tap water (plus 50 mg 13C-sodium acetate) given via nasogastric tube
  Interventions: Dietary Supplement: 75 g Erythritol; Other: 50 mg 13C-sodium acetate
- 75 g Glucose (Placebo Comparator): 75 g Glucose in 300 mL tap water (plus 50 mg 13C-sodium acetate) given via nasogastric tube
  Interventions: Dietary Supplement: 75 g Glucose; Other: 50 mg 13C-sodium acetate
- Tap water (Placebo Comparator): 300 mL tap water (plus 50 mg 13C-sodium acetate) given via nasogastric tube
  Interventions: Dietary Supplement: 300 mL tap water; Other: 50 mg 13C-sodium acetate

INTERVENTIONS:
Dietary Supplement: 0.52 g L-Tryptophan
  Arms: 0.52 g L-Tryptophan
Dietary Supplement: 1.56 g L-Tryptophan
  Arms: 1.56 g L-Tryptophan
Dietary Supplement: 1.56 g L-Leucine
  Arms: 1.56 g L-Leucine
Dietary Supplement: 50 g Xylitol
  Arms: 50 g Xylitol
Dietary Supplement: 75 g Erythritol
  Arms: 75 g Erythritol
Dietary Supplement: 75 g Glucose
  Arms: 75 g Glucose
Dietary Supplement: 300 mL tap water
  Arms: Tap water
Other: 50 mg 13C-sodium acetate

SUMMARY:
With this study the investigators investigate the effects of amino acids (tryptophan in two different concentrations, leucin) and sugar alcohols (xylitol, erythritol) on satiety mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal weight subjects with a body-mass index of 19.0-24.9
* Healthy obese subjects with a body-mass index of > 30
* Normal eating habits (no diets; no dietary changes; no special dietary habits, such as vegetarian/vegan)
* Age 18-40 years
* Stable body weight for at least three months

Exclusion Criteria:

* Smoking
* Substance abuse
* Regular intake of medications (except for oral contraceptives)
* Medical or psychiatric illness
* History of gastrointestinal disorders
* Food allergies
* Pregnancy, breast feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Effect of different aminoacids and sugar alcohols on secretion of satiation hormones | changes from baseline to three hours after treatment
  Plasma concentrations of glucose
Effect of different aminoacids and sugar alcohols on secretion of satiation hormones | changes from baseline to three hours after treatment
  Plasma concentrations of insulin are measured
Effect of different aminoacids and sugar alcohols on secretion of satiation hormones | changes from baseline to three hours after treatment
  Plasma concentrations of glucagon are measured
Effect of different aminoacids and sugar alcohols on secretion of satiation hormones | changes from baseline to three hours after treatment
  Plasma concentrations of glucagon-like Peptide (GLP-1) are measured
Effect of different aminoacids and sugar alcohols on secretion of satiation hormones | changes from baseline to three hours after treatment
  Plasma concentrations of PYY are measured
Effect of different aminoacids and sugar alcohols on secretion of satiation hormones | changes from baseline to three hours after treatment
  Plasma concentrations of cholecystokinin are measured

SECONDARY OUTCOMES:
Effect of different aminoacids and sugar alcohols on gastric emptying | changes from baseline to four hours after treatment
  measured by C13 breath test

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Phase 1 Research Unit, Basel, Switzerland

REFERENCES:
- [Derived] Meyer-Gerspach AC, Hafliger S, Meili J, Doody A, Rehfeld JF, Drewe J, Beglinger C, Wolnerhanssen B. Effect of L-Tryptophan and L-Leucine on Gut Hormone Secretion, Appetite Feelings and Gastric Emptying Rates in Lean and Non-Diabetic Obese Participants: A Randomized, Double-Blind, Parallel-Group Trial. PLoS One. 2016 Nov 22;11(11):e0166758. doi: 10.1371/journal.pone.0166758. eCollection 2016. PMID 27875537